CLINICAL TRIAL: NCT05310500
Title: Comparative Evaluation of Impact of Sodium Hypochlorite on Physical Properties of Finishing Files of ProTaper Gold And Dia-x ProTaper An In-Vitro Randomized Control Trial.
Brief Title: Comparative Evaluation of Impact of Sodium Hypochlorite on the Physical Properties of Protaper Gold and Dia-X ProTaper.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Iqra Kamal, Lecturer/ MDS Post graduate trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Iqrakamal01
Record Dates: First submitted 2021-12-08; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Dental Pulp Diseases
Keywords: root canal; pro taper gold; dia x pro taper; sodium hypochlorite
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ProTaper Gold (F2) - NaOCL (Experimental): ProTaper Files without NaOCL
  Interventions: Diagnostic Test: Finishing files of ProTaper Gold (F2) without effect to NaOCL
- ProTaper Gold (F2) + NaOCL (Experimental): ProTaper Files with NaOCL
  Interventions: Diagnostic Test: Finishing files of ProTaper Gold (F2) with effect to NaOCL
- Dia-X ProTaper (D4) - NaOCL (Experimental): Dia-X ProTaper (D4) without NaOCL
  Interventions: Diagnostic Test: Finishing files of Dia-X ProTaper (D4) without effect to NaOCL
- Dia-X ProTaper (D4) + NaOCL (Experimental): Dia-X ProTaper (D4) with NaOCL
  Interventions: Diagnostic Test: Finishing files of Dia-X ProTaper (D4) with effect to NaOCL

INTERVENTIONS:
Diagnostic Test: Finishing files of ProTaper Gold (F2) without effect to NaOCL — Finishing files of ProTaper Gold (F2) without effect to NaOCL
  Arms: ProTaper Gold (F2) - NaOCL
Diagnostic Test: Finishing files of ProTaper Gold (F2) with effect to NaOCL — Finishing files of ProTaper Gold (F2) with effect to NaOCL
  Arms: ProTaper Gold (F2) + NaOCL
Diagnostic Test: Finishing files of Dia-X ProTaper (D4) without effect to NaOCL — Finishing files of Dia-X ProTaper (D4) without effect to NaOCL
  Arms: Dia-X ProTaper (D4) - NaOCL
Diagnostic Test: Finishing files of Dia-X ProTaper (D4) with effect to NaOCL — Finishing files of Dia-X ProTaper (D4) without effect to NaOCL
  Arms: Dia-X ProTaper (D4) + NaOCL

SUMMARY:
The goal of the endodontic treatment is to make the root canal system free of the bacteria and its products to maximum extent, to allow healing of the inflamed apical periodontium.

Nickel titanium files have super elasticity, better cutting efficiency, and shapes canal anatomy more efficiently as compared to stainless steel manual files. Regardless of these properties, main shortcoming of Ni-Ti based files is their tendency to fracture unexpectedly inside the root canals. This abrupt file separation could be due to mechanical friction or chemical stimuli leading to the damage of surface contents (wear) and formation of micro cracks, waviness, scratches or roughness.

Sodium Hypochlorite is considered a gold standard irrigant in endodontics that renders bacteria free root canal system, but it has been postulated to have many shortcomings and certain concentrations of Sodium Hypochlorite affects the properties of Ni-Ti rotary instruments.

This clinical trial aimed to compare the physical properties (dimensional stability, deformation, surface roughness and metal slivering) and impact of 5.25% sodium hypochlorite on these physical properties of Protaper Gold finishing F2 Files and Dia-X ProTaper finishing D4 files when subjected to root canal preparation.

DETAILED DESCRIPTION:
It is estimated that over 95% of the reported cases of orofacial pain arises due to diseases of teeth and their associated supporting structures . There are several known etiological factors amongst which caries is the major cause of pulpal inflammation. The severity of the pulpal inflammation increases as the carious lesions progress deep into dentine and towards the pulp. This inflammatory process if left untreated triggers a cascade of events that leads to development of local or systematic pathologies. To resolve the symptoms of pulpitis, it becomes mandatory to carry out endodontic treatment by means of root canal treatment.

Root canal treatment is defined as "eradication and/or inhibition of apical periodontitis. Endodontic therapy is rendered as one of the most widely performed dental procedure as per survey conducted by AAE in 2007, the results showed the estimate of about 15.1 million RCT being performed annually in America.

Endodontic therapy is a categorization of treatment steps to eradicate the pulpal and Periapical infection from infected tooth. The therapy aims to decontaminate the tooth so that microbial invasion in future can be prevented. In case of already established Periapical lesion, root canal treatment facilitates healing of Periapical pathology, thus restoring the function of the dentition and at same time prevent reinfection of the tooth.

In order to carry out endodontic therapy successfully, the eradication of organic and inorganic debris from root canal system by means proper cleaning and shaping using chemo-mechanical debridement is compulsory. Adequate cleaning, shaping, proper irrigation and sealing of root canal is the triad for effective root canal therapy. The cleansing of the root canals is completed with the aid of endodontic files and irrigants, and later appropriate closing of the root canals by means of endodontic obturation is done.

The model of the germ theory of disease integrated with the development of dentistry had a direct effect on the practice of endodontics during the latter half of the 19TH century. The period between 1859 strengthened the importance of irrigation in endodontics when the use of syringes became frequent to remove "irritants" from root canal system and it was recommended by Taft until the mid-1940s when endodontics turn out to be a special field within dentistry and the American Endodontic Society was recognized.

An endodontic treatment comprises of removal of the microbes, flushes away loose, necrotic, contaminated elements from root canal system during the process of shaping of root canal. It is currently considered to be the best method to abolish dentine debris and tissue remnants during instrumentation of root canal system. Flushing of root canal also provides gross debridement, destruction of microbes, lubrication, dissolution of tissues and smear layer removal but the presence of anatomic variations particularly morphologic anomalies such as lateral canals, apical deltas, ramifications, and the thorough debridement of the root canal system has turn out to be a true clinical challenge in endodontics. Hence, root-canal preparation is important and also demanding for the clinician so as to ensure the longevity and success of root canal treatment.

There are three main issues that are at present considered to be most controversial and challenging in root canal shaping:

* To identify, Assess and enlarge the canals and avoiding the procedural errors.
* To establish and maintain the suitable working lengths during the course of the shaping of root canals.
* To select the size of preparation that permits sufficient disinfection and subsequent obturation.

Disinfection of entire root canal system is the key objective in root canal treatment and it may be achieved with mechanical instrumentation and chemical irrigation and with combination of intra- canal medicaments between treatment sessions.

In order to facilitate an adequate irrigation, several irrigant solutions have been formulated, tested and advocated but Sodium hypochlorite is well-thought-out as gold standard irrigant. Irrigants possess many advantages. Sodium Hypochlorite have tissue dissolving and anti-bacterial properties due to which it is widely used irrigant in root canal preparation but sodium hypochlorite also has some disadvantages like varying the mechanical properties of root dentine i.e. reduction in thickness, modulus of elasticity and flexural strength due to which the resistance to fracture of endodontic rotary instruments is altered . Sodium hypochlorite causes corrosion of metals also. The pattern of corrosion is such that it causes micro pitting by removing nickel from the surface. There is constant interaction of endodontic files with the sodium hypochlorite irrigant during instrumentation or disinfection procedure. Even immediate or short-duration interaction of this irrigant leads to alteration in the surface of Ni-Ti endodontic instruments.

The several reasons for the failure of endodontic treatment could be broadly classified into tooth-related factors and treatment-related factors. The tooth related factors include poor access, complex anatomy e.g. apical ramification, missed canals, accessory canals, insufficient cleaning and shaping of the root canal system and poor obturation. Treatment related factors are the procedural accidents for instance, instrument separation, ledge formation and perforation, hypochlorite accident etc. Unexpected ﬁle fracture is one of the main shortcomings of the several engines driven Ni-Ti endodontic instruments. Literature presents several studies that has shown the increased likelihood of file separation in apical third of root canal and that the finishing files are more prone to fracture as compared to shaping files. In order to reduce such problems, several changes in the manufacturing of Ni-Ti alloy has been carried out to enhance the super-elasticity of these instrument. Ni-Ti alloys are being thermally heat treated to enhance their consistency and efficacy to carry out endodontic preparation in curved canals as to reduce the fatigue stress and enhance the fracture resistance.

Various filing systems have been introduced, one of the novel system introduced as newer generation endodontic Ni-Ti Rotary system is ProTaper Gold Rotary filing System and another similar system is Dia-X ProTaper Rotary filing system. Literature suggests that these both systems are thermally heat-treated, files exhibit a convex triangular cross-section and continuous taper and offer more flexibility and increase in cyclic fatigue resistance with advancement in the metallurgy. In spite of many advantages, the frequency of file breakage during clinical use is very common.

Although several in-vivo & in-vitro studies have been carried to assess the different rotary Ni-Ti filing systems and many previous studies have been carried out to look for impact of Sodium hypochlorite irrigant on endodontic files leading to changes in the surface roughness, reduced resistance to fatigue, deformation and metal slivering. The aim of the study is to provide information about the impact of Sodium Hypochlorite irrigant at a standard concentration of 5.25% on the physical properties (dimensional stability, deformation, surface roughness and metal slivering) of Protaper Gold finishing F2 File and Dia-X ProTaper finishing D4 file when subjected to root canal preparation.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular first permanent molars
* A degree of root canal curvature ranging from 10 to 20 degree taper.

Exclusion Criteria:

* Teeth with internal and external resorption
* Teeth with calcified canals
* Previously endodontic treated teeth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Stereomicroscope and Optical microscope used to evaluate the changes of finishing files of ProTaper Gold (F2) and Dia-X ProTaper (D4). | 9 Months
  The change in dimensional stability of two file systems before and after clinical application and after exposure to Sodium Hypochlorite in root canal system.
Stereomicroscope and Optical microscope used to evaluate the changes of finishing files of ProTaper Gold (F2) and Dia-X ProTaper (D4). | 9 months.
  The change in surface roughness of two file systems before and after clinical application and after exposure to Sodium Hypochlorite in root canal system.
Stereomicroscope and Optical microscope used to evaluate the changes of finishing files of ProTaper Gold (F2) and Dia-X ProTaper (D4). | 9 months
  The change in Deformation of two file systems before and after clinical application and after exposure to Sodium Hypochlorite in root canal system.
Stereomicroscope and Optical microscope used to evaluate monitor the changes of finishing files of ProTaper Gold (F2) and Dia-X ProTaper (D4). | 9 months
  The Presence or absence of metal slivering of two file systems before and after clinical application and after exposure to Sodium Hypochlorite in root canal system.

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Kamal, BDS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow university of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zinelis S, Eliades T, Eliades G. A metallurgical characterization of ten endodontic Ni-Ti instruments: assessing the clinical relevance of shape memory and superelastic properties of Ni-Ti endodontic instruments. Int Endod J. 2010 Feb;43(2):125-34. doi: 10.1111/j.1365-2591.2009.01651.x. PMID 20078701

DOCUMENTS (1):
  • Informed Consent Form (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT05310500/ICF_000.pdf